CLINICAL TRIAL: NCT04940221
Title: Testing Informed Decision Making in Lung Cancer Screening
Acronym: TIDiL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: Thomas Jefferson University (Other); University of Delaware (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Heather Bittner Fagan, Physician - Family Medicine, Christiana Care Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 603913; U54GM104941 (NIH)
Record Dates: First submitted 2021-06-09; First posted 2021-06-25 (Actual); Results first posted 2022-10-20 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phone-delivered decision-counseling program for shared decision making in lung cancer screening (Experimental): All individuals who are eligible for lung cancer screening according to USPSTF criteria were invited to participate in the study and all patients who accepted the invitation and consented were slated to receive the intervention which was a phone-delivered on line decision-counseling program (DCP) and there was no one randomized or enrolled into a control group, nor was anyone randomized or enrolled into a usual care group.
  Interventions: Behavioral: Shared Decision Making

INTERVENTIONS:
Behavioral: Shared Decision Making — Telephone delivered non-persuasive shared decision-making for lung cancer screening.

SUMMARY:
Lung cancer screening rates are very low despite the fact that lung cancer screening could save many lives. People need to understand the risks and benefits to screening as well as their own beliefs about screening. This study builds an intervention in real world primary care that will help people make the right decision for them as well as help people to quit smoking. Interventions like this are needed to improve the screening rate and reduce death from lung cancer, which is the leading cancer killer.

DETAILED DESCRIPTION:
Lung cancer screening rates in the United States are very low- just 3.3% in 2010 and 3.9% in 2015. There is a critical need to develop and implement effective strategies to engage high-risk patients in a coordinated program of lung cancer screening, which includes shared-decision making. The investigators proposed to modify and expand a shared decision- counseling intervention previously developed in one primary care practice. The investigators measured lung cancer screening in our intervention group compared to a propensity-matched usual care cohort. The investigators compared patients recruited to patients who are not in order to identify potential sources of disparity in future work and the investigators developed a more intense smoking cessation component. Model interventions for shared-decision making in clinical practice are needed across a wide range of diseases and decisions.

ELIGIBILITY:
Inclusion Criteria:

* Current or former smoker
* Greater than or equal to 30 pack years smoking

Exclusion Criteria:

* Prior CT in last year
* Quit smoking greater than 15 years ago
* Current diagnosis of lung cancer

Ages: 55 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather B Fagan, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health System, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided
Pending data analytic support to de-identify data, will share entire study data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We identified 1359 individuals in our electronic medical record data who appeared to be current smokers within the age range of 55-78 years old. From this group, 1073 remained potentially eligible after chart review. From this group, 336 were reached by phone. From this group, 80 individuals were eligible and consented to be in our study.
Period: Overall Study
Arm/Group | Phone-delivered Decision-counseling Program for Shared Decision Making in Lung Cancer Screening
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phone-delivered Decision-counseling Program for Shared Decision Making in Lung Cancer Screening
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 66
  More than one race | 0
  Unknown or Not Reported | 0
pack-years [Mean (Standard Deviation); unit: (packs/day)*years] — It is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked.
  (packs/day)*years | 45.6 (16.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Received a Low Dose CT Scan of the Chest
Description: Percentage of individuals who have evidence of a low-dose CT scan of the chest in their electronic medical record at 1 year post intervention, as ascertained by chart audit by research assistance.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Phone-delivered Decision-counseling Program for Shared Decision Making in Lung Cancer Screening
Number analyzed (Participants) | 80
Participants | 18

ADVERSE EVENTS:
Time Frame: 1 year measured from the date of patient enrollment
Description: Serious adverse event, all-cause mortality, and other serious events were zero because lung cancer screening is part of standard clinical care. There were no adverse events within the course of this study.
Arm/Group | Phone-delivered Decision-counseling Program for Shared Decision Making in Lung Cancer Screening
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-08-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT04940221/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT04940221/ICF_001.pdf